CLINICAL TRIAL: NCT02488564
Title: Clinical and Translational Phase II Study of Liposomal Doxorubicin Plus Docetaxel and Trastuzumab with Metformin As Primary Systemic Therapy for Operable and Locally Advanced Recombinant Human ErbB-2 (HER2) Positive Breast Cancer
Brief Title: A Study of Liposomal Doxorubicin+Docetaxel+Trastuzumab+Metformin in Operable and Locally Advanced HER2 Positive Breast Cancer
Acronym: met-HEReMYTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST174.09
Record Dates: First submitted 2015-06-17; First posted 2015-07-02 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: HER-2 Positive Breast Cancer
Keywords: HER-2 Positive Breast Cancer; operable breast cancer; locally advanced breast cancer; no prior therapy; pCR
MeSH Terms: interventions — liposomal doxorubicin; Doxorubicin; Docetaxel; Trastuzumab; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liposomal doxorubicin +Docetaxel+Trastuzumab+Metformin (Experimental): Day 1: Liposome-encapsulated doxorubicin, 50 mg/m2 IV 1 hour infusion; Day 2 and 9: Docetaxel, 30 mg/m2 IV 1 hour infusion; Day 2, 9 and 16: Trastuzumab 4 mg/kg for the first infusion loading dose, then 2 mg/kg/week for subsequent injections.
  Day -13 to 0: Metformin is administered as single agent. From day -13 to day -11, Metformin 1000 mg will be administered once a day; from day -10 Metformin 1000 mg will be administered twice a day continuously until end of the study treatment.
  Interventions: Drug: Liposomal doxorubicin; Drug: Docetaxel; Drug: Trastuzumab; Drug: Metformin

INTERVENTIONS:
Drug: Liposomal doxorubicin — 50 mg/m2 by intravenous infusion over a period of 1 hour on day 1 of each cycle repeated every 21 days. A final concentration of between 0.4 to 1.2 mg/ml doxorubicin hydrochloride, is required
  Other Names: Myocet®
Drug: Docetaxel — 30 mg/m2 by intravenous infusion over a period of 1 hour on day 2 and 9, every 3 week.They will be given for 6 cycles.
  Other Names: taxotere
Drug: Trastuzumab — 4 mg/kg for the first administration (day 2 cycle 1) and 2 mg/kg for subsequent administrations. Trastuzumab will be given weekly for the duration of chemotherapy (day 2, 9, 16), then will be administered at the dose of 6 mg/Kg every 3 weeks until completion of 52 weeks of treatment.
  Other Names: herceptin
Drug: Metformin — It is administered as single agent from day -13 to 0. From day -13 to day -11, Metformin 1000 mg will be administered once a day; from day -10, Metformin 1000 mg will be administered twice a day continuously until end of the study treatment.

SUMMARY:
It is a multicenter, open-label, two stage phase II trial, to assess activity, safety and potential early predictors of response in neoadjuvant setting. Patients with operable breast cancer (T1c and cytologically N1-2, or cT2-3, N0-N2, M0) or locally advanced breast cancer (T4a-d, N0-N2, M0) with overexpression or amplification of HER2 (AJCC 7th edition 2010) are included in the study.

The primary objective is to evaluate the pathological complete response rate (pCR).

The secondary objectives are:

* to evaluate the clinical response rate (RR).
* to evaluate the feasibility and systemic tolerance, with particular attention to cardiac toxicity.
* to evaluate the conservative surgery rate.

Total duration of the trial is 36 months; planned treatment are 6 cycles of chemotherapy. At every cycle (every 21 days) will be administered:

Day 1: Liposome-encapsulated doxorubicin, 50 mg/m2 IV 1 hour infusion; Day 2 and 9: Docetaxel, 30 mg/m2 IV 1 hour infusion; Day 2, 9 and 16: Trastuzumab 4 mg/kg for the first infusion loading dose, then 2 mg/kg/week for subsequent injections. Day -13 to 0: Metformin is administered as single agent. From day -13 to day -11, Metformin 1000 mg will be administered once a day; from day -10 Metformin 1000 mg will be administered twice a day continuously until end of the study treatment.

DETAILED DESCRIPTION:
Multi-center, open-label phase II trial to assess activity of this chemotherapy scheme evaluated by pathologic complete response rate (pCR).

Planned treatment are 6 cycles of chemotherapy.

At every cycle (every 21 days) will be administered:

Day 1: Liposome-encapsulated doxorubicin, 50 mg/m2 IV 1 hour infusion; Day 2 and 9: Docetaxel, 30 mg/m2 IV 1 hour infusion; Day 2, 9 and 16: Trastuzumab 4 mg/kg for the first infusion loading dose, then 2 mg/kg/week for subsequent injections Day -13 to 0: Metformin is administered as single agent. From day -13 to day -11, Metformin 1000 mg will be administered once a day; from day -10 Metformin 1000 mg will be administered twice a day continuously until end of the study treatment.

Total duration of the trial: 36 months Enrollment period: 24 months Treatment: maximum of 6 cycles (5 months) per patient Follow-up for recurrence: every six months for 5 years, than once a year until 10 years after surgery.It's necessary to recruit 46 patients for clinical objectives evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed breast cancer
* HER2 overexpressing cancer
* Patients with operable breast cancer (T1c and cytologically N1-2, or cT2-3, N0-N2, M0) or locally advanced breast cancer (T4a-d, N0-N2, M0) (AJCC 7th edition 2010).
* No prior therapy for breast cancer
* Both sexes, age ≥ 18 years and < 75 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Life expectancy > 3 months
* Neutrophil count ≥ 2 x 109/ L, leukocytes count ≥ 3 x 109/ L and platelet count ≥ 100 x 109/ L
* Total bilirubin ≤ 1 upper-normal limits (UNL) of the Institutional normal values and alanine aminotransferase (ASAT (GOT) and/or alanine aminotransferase ALAT (GPT) ≤ 2.5 UNL, alkaline phosphatase ≤ 5 UNL. Patients with ASAT and/or ALAT > 1.5 UNL and alkaline phosphatase > 2.5 UNL aren't eligible for the trial.
* Creatinine ≤ 1.5 mg/dL
* Left ventricular ejection fraction (LVEF) ≥ 50% (evaluated by echocardiogram or multiple gated acquisition scan (MUGA) scan -only one method must be employed for each patient)
* Written informed consent
* Homa Index calculated using the Matthews'formula

EXCLUSION CRITERIA:

* Prior chemotherapy or radiotherapy for breast cancer.
* History of prior malignancy in the last 10 years (other than non-melanoma skin cancer or excised cervical carcinoma in situ).
* Other serious illness or medical condition
* Congestive heart failure or angina pectoris even if medically controlled. Previous history of myocardial infarction, uncontrolled high risk hypertension or arrhythmia
* History of significant neurologic or psychiatric disorders including dementia or seizures
* Active infection
* Concurrent treatment with other experimental drugs.
* Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
* Geographic inaccessibility to treatment and followup
* Pregnant and lactating women
* Diabetes-insulin dependant and non-insulin dependant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response rate(pCR) | up to 36 months
  Complete pathologic response will be defined as no invasive residuals in breast and axillary nodes. In situ tumor residuals are considered as complete response rate

SECONDARY OUTCOMES:
clinical response rate (RR) | up to 36 months
  The clinical response rate (RR) will be including Pathological Complete Response, Clinical Complete Response and Clinical Partial Response (Response Evaluation Criteria in Solid Tumors (RECIST) criteria).
evaluation of toxicity | up to 36 months
  All patients will be evaluable for toxicity from the time of their first treatment with Metformine. The toxicity will be recorded according to the CTC-AE, version 4.0 in the safety population until Follow-up is completed (36 months)
conservative surgery rate | up to 36 months
  evaluation of the number of patients who underwent conservative surgery

CONTACTS AND LOCATIONS:
Overall Officials: Anna Fedeli, MD, Principal Investigator — IRST IRCCS, Meldola-Cesena
Locations (9):
- Italy (9):
  - IRST Oncologia medica, Meldola, FC
  - Oncologia Medica AOU Ferrara, Ferrara, FE
  - Oncologia Medica, Policlinico di Modena, Modena, MO
  - Oncologia Medica Ospedale Guglielmo da Saliceto, Piacenza, PC
  - Oncologia , IRCCS azienda ospedaliera S.Maria Nuova, Reggio Emilia, RE
  - U.O Oncologia AUSLdella Romagna, Rimini, RN
  - Day Hospital Oncologico, Ospedale Guastalla, Guastalla
  - Oncologia Medica AUSL Imola, Imola
  - Oncologia Medica AOU Parma, Parma